

*Title:* A Placebo-controlled, Randomized, Double-masked, Cross-over Acute Intervention Study Investigating the Effects of Cocoa Flavanols on Peripheral Endothelial Function in the Context of Prolonged Sitting in Healthy Older Adults

Protocol ID/ Ethics ID: ERN\_19-0851B

Date of Approval: 14th September 2021



## School of Sport, Exercise and Rehabilitation Sciences

## Participant Consent Form

| Study Title: | The impact of cocoa flavanols on blood vessel function during uninterrupted sitting in older adults | | |
|---|---|---|---|
| Investigators: | Dr Catarina Rendeiro, Dr Sam Lucas, Mr Alessio Daniele, and Prof Carolyn Greig | | |
| Name: | Date of Birth: | | |
| Address: | Telephone: | | |
| Please read the | statements carefully | and initial the bo | oxes if you agree. |
| | _ | | sed the experiment with one of procedures to my satisfaction. |
| I understand that I am volunteering to participate in the experiment by my choice and that I may stop and withdraw from the experiment at any time. | | | |
| I confirm that I have not been treated for any cardiovascular, metabolic, neurological, or respiratory conditions in the past. | | | |
| I confirm that I do not have any food allergies to the best of my knowledge | | | |
| I understand that the data collected during the study may be looked at by responsible individuals from the University of Birmingham where it is relevant to my taking part in this research. I give permission for these individuals to have access to my data and understand that any information will be kept strictly confidential. | | | |
| I understand that my digital data will be stored for a minimum of 10 years in accordance with University of Birmingham policies on password protected systems accessible only to research personnel associated with this study. I agree to this. | | | |
| I understand that my questionnaire data will be stored for a minimum of 10 years in accordance with University of Birmingham policies in a locked cabinet only accessible to the research personnel associated with this study. I agree to this. | | | |
| I would like to receive a summary of the study findings (tick $\checkmark$ your response) YES $\square$ NO $\square$ | | | |
| I agree to the arrangements described in the Information Sheet as they relate to my participation. Then, I agree to participate in this study. | | | |
| Name of the Pa | articipant (PRINT) | Date | Signature |
| Name of the Re | esearcher (PRINT) | Date | Signature |